CLINICAL TRIAL: NCT04535024
Title: Phase II Trial of Multisite Stereotactic Ablative Radiotherapy (SABR) Combined With Sintilimab for Microsatellite Stable (MSS) Oligometastatic Colorectal Cancer
Brief Title: The Combination of Immunotherapy and Stereotactic Ablative Radiotherapy in MSS Oligometastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2019-251-1881
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A total of 60 MSS oligometastatic colorectal cancer patients will receive multisite SABR followed by Sintilimab within one week from completion.
  The dosing will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR); Drug: Sintilimab

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — We plan to irradiate as many metastatic lesions as possible, in the precondition that normal tissues can tolerate.
  Target dose will be adjusted depending on site of the lesion and organs at risk (BED > 100Gy).
  Treatment schedule is once per day and five days per week. Sequence of irradiation for multiple metastases is at the discretion of the investigators based on their experience.
Drug: Sintilimab — Starts within one week upon SABR completion: 200mg, d1, q3w; Continued until disease progression, unacceptable toxicity or patient withdrawal.

SUMMARY:
This is a prospective, single-center, single-arm phase II clinical trial. This study aims to evaluate the safety and tolerability of stereotactic ablative radiotherapy (SABR) in combination with Sintilimab, and to examine the impact of the combination therapy on tumor control, long-term survival and quality of life in patients with microsatellite stable (MSS) oligometastatic colorectal cancer.

A total of 60 MSS oligometastatic colorectal cancer patients will be recruited and receive multisite SABR followed by immunotherapy of Sintilimab within one week from completion. Sintilimab will be given at a fixed dose of 200mg (100mg if weight < 50 kg) via intravenous infusion on the first day of each cycle, repeated every three weeks. The dosing will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal. The tumor regression, disease control, adverse events and long-term survival will be analyzed.

DETAILED DESCRIPTION:
Immune-checkpoint inhibitor (ICI) has led to a paradigm shift in the treatment of patients with metastatic cancer, as proved by improved survival and durable responses in a group of these patients. However, the response rates to ICI when given alone are limited. In gastrointestinal cancer, patients with microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors shown a response rate of approximately 40% to ICI, while patients with microsatellite stable (MSS) or mismatch repair-proficient (pMMR) tumors respond poorly to ICI. Such observations have spurred efforts to expand the benefit of immunotherapy, especially in these immune "non-sensitive" tumors, by combining ICI with treatments that induce T-cell associated immune response such stereotactic ablative radiotherapy (SABR).

High-dose ablative radiation was showed to facilitate immunotherapy through promote the activation of innate and adaptive immune responses against tumors in preclinical model and early phase clinical trials. However, a large portion of trials which were launched to test the efficacy of radiotherapy and immunotherapy produced suboptimal results. One important reason could be that majority of these trails were designed with single lesion irradiation, which is insufficient to unveil enough tumor antigens and/or to break the barrier of immunosuppressive tumor microenvironment (TME).

The investigators hypothesized that irradiation to multiple or all sites of diseases is more likely to produce an optimized regimen with ICI by broadly stimulate anti-tumor immunity and reduce tumor burden. Therefore, this study plans to administrate SABR to as many metastatic lesions as possible, in combination with ICI (Sintilimab) in patients with MSS oligometastatic colorectal cancers, to assess safety and tolerability of the regimen, and evaluate its early efficacy as well.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old, regardless of gender
* Fully informed and willing to provide written informed consent for the trial
* ECOG performance status 0-1
* Has an investigator determined life expectancy of at least 6 months
* Histologically confirmed colorectal adenocarcinoma, with MSS or pMMR status
* Has 2-5 measurable metastatic lesions detected on imaging, with none of them indicated for surgery; or the participant refuses to receive surgery. Biopsy of metastasis is preferred, but not required
* Has undergone at least one dose of first-line systemic chemotherapy, except for any type of immunotherapy
* Multiple sites of lesions can be safely treated by SABR, and at least one lesion spared from irradiation, so as for assessment. The maximum diameter of each lesion for irradiation is no more than 5cm.
* Demonstrate adequate organ function
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Pregnant or lactating women
* Serious medical comorbidities precluding radiotherapy
* Prior radiotherapy to a site requiring treatment
* Malignant pleural effusion
* Inability to treat all sites of active disease
* Has clinical or radiologic evidence of spinal cord compression or tumor within 3mm of spinal cord on MRI.
* Dominant brain metastasis requiring surgical decompression
* Has prior treatment with cancer immunotherapy including, but not limited to immune checkpoint inhibitors.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10 mg Prednisone daily or equivalent at time of trial treatment.
* Has a known history of active Bacillus Tuberculosis
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Hypersensitivity to PD-1 inhibitor or any of its excipients.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered from adverse events due to a previously administered agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years
  The percentage of patients with objective response in the non-irradiated metastatic lesions. Objective response is defined as complete response (CR) or partial response (PR) per response evaluation criteria (RECIST v1.1) and the immune related response criteria (iRECIST) after treatment.

SECONDARY OUTCOMES:
Disease Control Rate | Up to 2 years
  The percentage of patients with disease control in the non-irradiated metastatic lesions. Disease control is defined as CR, PR, or stable disease (SD) per RECIST v1.1 and iRECIST after treatment.
Duration of Response | Up to 2 years
  Defined as the time between PR/CR and subsequent progression disease (PD) per RECIST v1.1 and iRECIST or death from any cause.
Progression-Free Survival | Up to 3 years
  Defined as the time from initiation of treatment to PD or death from any cause.
Overall Survival | Up to 3 years
  Defined as the time from initiation of treatment to death from any cause.
Acute Toxicity | Up to 2 years
  The percentage of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China